CLINICAL TRIAL: NCT02011152
Title: The Effect of Intravenous Magnesium Sulfate Infusion on Sensory Spinal Block and Postoperative Pain Score in Abdominal Hysterectomy
Brief Title: Spinal Anesthesia Magnesium Infusion
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Fatih Kahraman, The effect of intravenous magnesium sulfate infusion on sensory spinal block and postoperative pain score in abdominal hysterectomy, Karadeniz Technical University
Other Study IDs: 199812; spinal magnesium (Other: spinal)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Operation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to investigate the effect of i.v. infusion of magnesium sulphate during spinal anesthesia on duration of spinal block and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II, aged between 18 and 65 female patients undergoing abdominal hysterectomy

Exclusion Criteria:

* severe cardiovascular, renal and hepatic dysfunction, neuromuscular diseases, using calcium channel blockers, and inappropriate for spinal anesthesia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 and 65 female patients undergoing abdominal hysterectomy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 1998-12; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
pain scores | 6 mo

SECONDARY OUTCOMES:
sensory block | 6 mo

OTHER OUTCOMES:
motor block | 6mo

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Kahraman, Principal Investigator — KTU